CLINICAL TRIAL: NCT04477707
Title: Observational Study of Routine Ophthalmological Examinations of Patients Included in the 2 Bayer Sponsored Phase 3 Clinical Trials FIDELIO and FIGARO to Investigate the Effect of Finerenone on Delaying the Progression of Diabetic Retinopathy
Brief Title: A Study That Uses Data From Routine Eye Examinations of Patients Participating in Studies FIDELIO-DKD and FIGARO-DKD to Explore Whether Finerenone Can Delay the Progression of a Diabetes Complication That Affects the Eyes (Diabetic Retinopathy ,DR)
Acronym: ReFineDR
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21311
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group: Patients received treatment in phase 3 clinical trials FIDELIO or FIGARO.
  Interventions: Drug: Finerenone (BAY94-8862)
- Placebo group: Patients received placebo in phase 3 clinical trials FIDELIO or FIGARO.

INTERVENTIONS:
Drug: Finerenone (BAY94-8862) — 10 mg or 20 mg Finerenone tablet to be given orally, once daily, administered in the FIDELIO or FIGARO clinical trial.
  Groups: Treatment group

SUMMARY:
Diabetic retinopathy (DR) is a diabetes complication caused by damage to the small blood vessels inside the retina at the back of the eye. Diabetic retinopathy may cause mild vision problems or eventually blindness. Diabetes is a condition that makes your blood sugar levels higher than they should be.

In the early stages of diabetic retinopathy - called non-proliferative diabetic retinopathy (NPDR)- increased blood sugar levels lead to damage to the tiny blood vessels of the retina. This damage results in small outpouchings of the vessel lumens leading to rupture. At the same time the blood vessels can leak and making the retina swell and can cause so called macula edema. In these early stages of DR current treatment to reduce the risk of this eye complication is focused on controlling blood sugar levels and blood pressure.

Participants in this study have NPDR, Type 2 Diabetes (T2D) and Chronic Kidney Disease (CKD), a condition in which the kidneys become damaged and do not work as they should. These participants are already taking part in one of the phase 3 studies (FIDELIO-DKD and FIGARO-DKD). They study the effect of Finerenone on delaying kidney disease progression and reducing the risk of events that may cause damage to the heart and blood vessels To learn more about the effect of Finerenone on diabetic retinopathy, data from routine eye examinations performed during the two phase 3 studies will be collected and analyzed. All male and female participants included in this study are at least 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in ReFineDR
* Included in FIDELIO or FIGARO, and with DR as medical history
* Documented NPDR in at least one eye, as documented by ophthalmological records within 6 months prior to baseline in FIDELIO or FIGARO, and up to one month after baseline in FIDELIO or FIGARO
* An ophthalmological assessment available 6 month before or maximum 1 month after the baseline examination in FIDELIO or FIGARO, and at least one additional assessment afterwards.

Exclusion Criteria:

* Patients with PDR, macular edema or anterior segment complications present at baseline in FIDELIO or FIGARO in at least one eye.
* Patients with any documentation of prior or planned retinal laser treatment, intravitreal injection or vitrectomy at baseline in FIDELIO or FIGARO in at least one eye.
* Patients with any other retinal disease documented at baseline in FIDELIO or FIGARO in at least one eye that would likely interfere with the study objectives (e.g. neovascular age-related macular degeneration or retinal vein occlusion).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of patients included in FIDELIO or FIGARO with NPDR. Patients with at least one routine ophthalmological assessment available at baseline in FIDELIO or FIGARO, and one additional measurement at a later time point.
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Progression of non-proliferative diabetic retinopathy (NPDR) | After start of treatment until end of Year 2
  Progression of non-proliferative diabetic retinopathy (NPDR) defined by the occurrence of vision-threatening events i.e. proliferative diabetic retinopathy (PDR), diabetic macular edema (DME), anterior segment neovascularization (ASN) until the end of Year 2 after start of treatment

SECONDARY OUTCOMES:
Progression of non-proliferative diabetic retinopathy (NPDR) | After start of treatment until end of Year 1
  Progression of non-proliferative diabetic retinopathy (NPDR) defined by the occurrence of vision-threatening events i.e. proliferative diabetic retinopathy (PDR), diabetic macular edema (DME), anterior segment neovascularization (ASN) until the end of Year 1 after start of treatment
Progression of non-proliferative diabetic retinopathy (NPDR) to proliferative diabetic retinopathy (PDR) | After start of treatment until end of Year 1 and end of Year 2
Occurrence of diabetic macular edema (DME) | After start of treatment until end of Year 1 and end of Year 2
Occurrence of anterior segment neovascularization (ASN) | After start of treatment until end of Year 1 and end of Year 2
Change in severity of diabetic retinopathy (DR) | From strat of treatment to the end of Year 1 and end of Year 2

CONTACTS AND LOCATIONS:
Locations (62):
- United States (10):
  - California Institute of Renal Research - Chula Vista, Chula Vista, California
  - California Institute of Renal Research, Inc. - El Centro, El Centro, California
  - Elixia at Florida Kidney Physicians Southeast, Fort Lauderdale, Florida
  - John H Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Crescent City Clinical Research Center, LLC, Metairie, Louisiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Office of Osvaldo A. Brusco, MD, Corpus Christi, Texas
  - MedResearch, Inc., El Paso, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
- Argentina (5):
  - Centro Médico Viamonte, CABA, Buenos Aires
  - Centro de Investigación Médica Lanús, Lanús, Buenos Aires
  - Hospital Privado de la Comunidad, Mar del Plata, Buenos Aires
  - Investigación Clínica Aplicada, Ciudad Autón. de Buenos Aires, Ciudad Auton. de Buenos Aires
  - Salud renal, San Luis
- China (2):
  - Huai'an First People's Hospital, Nanjing Medical University, Huai'an, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical university, Nanjing, Jiangsu
- Centro de Diabetes Cardiovascular IPS Ltda., Barranquilla, Atlántico, Colombia
- Denmark (6):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Skejby, Aarhus N
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Holbæk Sygehus, Holbæk
  - Holstebro Hospital, Endocrinology dept., Holstebro
  - Viborg Sygehus, Viborg
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital Hong Kong, Shatin
- Israel (3):
  - Edith Wolfson Medical Center, Holon
  - Meir Medical Center, Kfar Saba
  - Clalit Health Services, Midgal Hamea, Tel Aviv
- Italy (2):
  - ASST Bergamo Ovest, Bergamo, Lombardy
  - ASL TO5, Turin, Piedmont
- Japan (9):
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Steel Memorial Yawata Hospital, Kitakyushu, Fukuoka
  - Hirohata Naika Clinic, Kitakyushu, Fukuoka
  - Medical corporation Yamagata Naika Clinic, Asahikawa, Hokkaido
  - Naka Kinen Clinic, Naka, Ibaraki
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa
  - Sasebo Chuo Hospital, Sasebo, Nagasaki
  - Fukui Prefectural Hospital, Fukui
  - Osaka General Medical Center, Osaka
- APDP, Lisbon, Portugal
- Russia (9):
  - First City Clinical Hospital n.a. E.E. Volosevich, Arkhangelsk
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - Krasnoyarsk Clinical Hospital n.a. N.S. Karpovich, Krasnoyarsk
  - PHI "Central Clinical Hospital "RZD-Medicine", Moscow
  - City Clinical Hospital #13 Nizhny Novgorod, Nizhny Novgorod
  - Novosibirsk State Medical University, Novosibirsk
  - Saratov City Clinical Hospital #9, Saratov
  - Voronezh Regional Clinical Consultancy-Diagnostic Center, Voronezh
  - City Outpatient Clinic #4, Voronezh
- South Korea (3):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Kangnam Sacred Heart Hospital, Seoul
- Spain (2):
  - Hospital SAS de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario Virgen de las Nieves|Medicina Interna, Granada
- Sweden (2):
  - Avdelningen för kliniska prövningar AKP, Örebro
  - Akademiska Sjukhuset Njurmottagningen, Uppsala
- Taiwan (5):
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/